CLINICAL TRIAL: NCT01466036
Title: An Open-Label, Phase II Study of Cabozantinib (XL184) in Advanced Pancreatic Neuroendocrine and Carcinoid Tumors
Brief Title: Cabozantinib in Advanced Pancreatic Neuroendocrine and Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-274
Record Dates: First submitted 2011-10-24; First posted 2011-11-07 (Estimated); Results first posted 2023-07-20 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Carcinoid Tumor; Pancreatic Neuroendocrine Tumor
Keywords: metastatic
MeSH Terms: conditions — Carcinoid Tumor; Adenoma, Islet Cell; Neoplasm Metastasis | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metastatic or Unresectable PNET (Experimental): An anticipated 35 patients with pancreatic neuroendocrine tumors receiving cabozantinib
  Interventions: Drug: Cabozantinib
- Metastatic or Unresectable Carcinoid (Experimental): An anticipated 35 patients with advanced or metastatic carcinoid tumor receiving cabozantinib
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — 60 mg QD orally in cycles of 28 days
  Other Names: XL184

SUMMARY:
Cabozantinib works by blocking the growth of new blood vessels that feed a tumor. In addition to blocking the formation of new blood cells in tumors, cabozantinib also blocks pathways that may be responsible for allowing cancers cells to become resistant to other "anti-angiogenic" drugs. Cabozantinib has been studied or is being study in research studies as a possible treatment for various types of cancer, including prostate cancer, brain cancer, thyroid cancer, lung cancer, and kidney cancer.

In this research study, the investigators wish to learn if cabozantinib is effective in treating patients with pancreatic neuroendocrine and carcinoid tumors.

DETAILED DESCRIPTION:
Subjects will take cabozantinib orally, once per day, in cycles of 28 days.

During each cycle subjects will have the following procedures:

* Physical examination, including measurement of weight and vital signs
* Questions regarding any side effects
* Blood sample (about 1 tablespoon) for routine laboratory tests of blood cell counts, blood chemistries, organ function and blood clotting
* Blood sample (about 4 tablespoons) for research test to measure biomarkers to assess the response to study drug
* Urine sample for routine urine tests to monitor health

On Day 15 (beginning of week 3) during the first 3 cycles:

* Physical examination, including measurement of weight and vital signs
* Questions regarding any side effects
* Blood sample (about 1 tablespoon) for routine laboratory tests of blood cell counts, blood chemistries, organ function and blood clotting
* Blood sample (about 4 tablespoons) for research test to measure biomarkers to assess the response to study drug Subjects will receive a CT scan or MRI every two cycles (every two months) to evaluate disease.

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic, histologically-confirmed, carcinoid or pancreatic neuroendocrine tumor. Tumors must be considered well- or moderately-differentiated. Patients with poorly differentiated neuroendocrine carcinoma or cell carcinoma are excluded from the study.
* A tumor sample is required for enrollment (except for patients diagnosed > 7 years ago).
* Must have measurable disease by RECIST criteria
* Must have evidence of progressive disease within 12 months of study entry
* Prior or concurrent therapy with somatostatin analogs is permitted. If on somatostatin/octreotide, must be on a stable dose for at least two months.
* Age ≥ 18 years
* No major surgery or radiation in the prior 4 weeks prior to enrollment
* No prior therapy with cabozantinib
* ECOG Performance status ≤ 1
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin </= 1.5X normal institutional limits
  * AST (SGOT) and ALT (SGPT) </=2.5x normal institutional limits, or < 5x if liver metastases are present
  * Creatinine </= 1.5x normal institutional limits or creatinine clearance > 50mL/min
  * Urine Protein:Creatinine ratio of <1
  * Lipase < 1.5X upper limit of normal
  * Serum Albumin ≥ 2.8 g/dl
* Sexually active subjects must agree to use medically accepted methods of birth control during the course of the study and for 3 months following discontinuation of study treatments (excluding women who are not of child bearing potential and men who have been sterilized).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Subjects receiving any other standard or investigational anticancer agents, with the exception of somatostatin/octreotide therapy. If patients has received prior cytotoxic chemotherapy, must be at least three weeks since last treatment before first dose of study treatment.
* Major surgery or radiation treatment <4 weeks prior to enrollment. In addition, cannot have received radiation to the thorax or gastrointestinal tract within three months of the first dose of study treatment.
* Cannot have received radionuclide treatment within 6 weeks of first dose of study treatment.
* High grade or poorly differentiated neuroendocrine tumors
* Ongoing immunosuppression with systemic steroids or other immune modulator
* Presence of CNS metastatic disease
* Uncontrolled hypertension defined by SBP > 140 or DBP > 90 despite titration of anti hypertensive medications
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements. Congestive heart failure or symptomatic coronary artery disease within 3 months prior to enrollment
* Cerebrovascular accident within prior 6 months
* The subject has a history of clinically significant hematemesis or a recent history of hemoptysis of > 2.5 mL of red blood or other signs indicative of pulmonary hemorrhage or evidence of endobronchial lesion(s).
* The subject has a pulmonary lesion abutting or encasing a major blood vessel.
* Previous history of pulmonary embolism or deep venous thrombosis
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or Coumadin-related agents, heparin, thrombin or FXa inhibitors, and antiplatelet agents (eg, clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic Low Molecular Weight Heparin (LMWH) are permitted.
* At the time of screening, active peptic ulcer disease or active inflammatory bowel disease (including ulcerative colitis or Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis, or appendicitis.
* History of abdominal fistula, gastrointestinal perforation, bowel obstruction, gastric outlet obstruction, or intra-abdominal abscess within six months of study enrollment.
* History of GI surgery within the past 28 days. If >28 days since GI surgery, must have confirmation of complete healing before initiating treatment with study drug.
* Other disorders associated with a high risk of fistula formation, including PEG tube placement within 3 months before the first dose of study therapy or concurrent evidence of intraluminal tumor involving the trachea or esophagus.
* Other clinically significant disorders such as:

  * Active infection requiring systemic treatment
  * Serious non-healing wound/ulcer/bone fracture
  * History of organ transplant
  * Concurrent uncompensated hypothyroidism or thyroid dysfunction
  * History of major surgery within 4 weeks or minor surgical procedures within one week before randomization
* The subject has a corrected QT interval calculated by the Fridericia formula > 500ms within 28 days before randomization.
* Severely impaired lung function
* Concurrent malignancy (other than non-melanoma skin cancer) diagnosed within the past 3 years or any currently active malignancy
* Pregnant women are excluded from this study due to the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with the treatment protocol, breastfeeding should be discontinued if the mother is treated on protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-07; Primary Completion 2021-08 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chan, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic or Unresectable PNET: patients with pancreatic neuroendocrine tumors receiving cabozantinib
  Cabozantinib: 60 mg QD orally in cycles of 28 days
- Metastatic or Unresectable Carcinoid: patients with advanced or metastatic carcinoid tumor receiving cabozantinib
  Cabozantinib: 60 mg QD orally in cycles of 28 days
Period: Overall Study
Arm/Group | Metastatic or Unresectable PNET | Metastatic or Unresectable Carcinoid
Started | 20 | 41
Completed (treatment was indefinite) | 0 | 0
Not Completed | 20 | 41
Not completed — Death | 1 | 1
Not completed — Physician Decision | 0 | 4
Not completed — Adverse Event | 2 | 6
Not completed — Withdrawal by Subject | 2 | 8
Not completed — progression/relapse | 14 | 21
Not completed — prolonged treatment delay | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metastatic or Unresectable PNET | Metastatic or Unresectable Carcinoid | Total
Number analyzed (Participants) | 20 | 41 | 61
Age, Continuous [Median (Full Range); unit: years] | 55 [42 to 79] | 63 [42 to 77] | 60 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 23 | 31
  Male | 12 | 18 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The objective response rate of cabozantinib was evaluated according to RECIST v 1.1 criteria (Response Evaluation Criteria In Solid Tumors v 1.1). Disease was assessed using CT and/or MRI scans. RECIST 1.1 criteria include the following categories of disease response: Complete Response (CR) = disappearance of all target lesions; Partial Response (PR) = 30% or more decrease in the sum of the longest diameter of target lesions; Stable disease (SD) = less than 30% decrease but no more than 20% increase in sum of the longest diameter of target lesions. Objective response rate consisted of CR + PR.
Time Frame: Imaging was performed cycles 2,4,6 every 8 weeks for the first 24 weeks, then every 3rd cycle every 12 weeks until progression or EOT. Median treatment duration was 8 cycles for the Carcinoid cohort and 12.5 cycles for the PNET cohort. Cycle=28 days.
Population: Response rate by RECIST 1.1 was calculated by including all patients who started study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic or Unresectable PNET | Metastatic or Unresectable Carcinoid
Number analyzed (Participants) | 20 | 41
Participants | 3 | 7

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival was defined as time in months from initiation of treatment until disease progression by RECIST 1.1 criteria or death from any cause. Progressive disease by RECIST 1.1 criteria is defined as at least a 20% increase in the sum of the longest dimensions of target lesions, taking as reference the smallest sum of longest dimensions recorded since the treatment started; the appearance of one or more new lesions; unequivocal progression of existing non-target lesions.
Time Frame: Restaging imaging was performed after cycles 2, 4, and 6 (every 8 weeks for the first 24 weeks), then every 3rd cycle (every 12 weeks) until disease progression or end of study treatment. Median follow-up is 89.1 months. Cycle = 28 days.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic or Unresectable PNET | Metastatic or Unresectable Carcinoid
Number analyzed (Participants) | 20 | 41
months | 21.1 [8.6 to 32.0] | 17.6 [8.3 to 23.8]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Median follow-up time of 89.1 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic or Unresectable PNET | Metastatic or Unresectable Carcinoid
Number analyzed (Participants) | 20 | 41
months | 37.3 [14.5 to 70.7] | 36.1 [20.6 to 65.5]

ADVERSE EVENTS:
Time Frame: Participants were followed for AEs and SAEs starting from the first dose of study treatment, throughout the study, and through 30 days from the last study treatment. Median treatment duration was 8 cycles for the Carcinoid cohort and 12.5 cycles for the PNET cohort. Patients were followed for AEs during the time on treatment plus 30 days (median of 9.6 months). Participants were followed for All-Cause Mortality for longer (median 89.1 months).
Description: Adverse Event (AE): An adverse event (AE) is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. Abnormal laboratory values or diagnostic test results constitute adverse events only if they are determined to be of clinical significance or require treatment or further diagnostic tests
Groups:
- Metastatic or Unresectable PNET: patients were stratified by primary tumor site but received the same treatment. This cohort had pancreatic neuroendocrine tumors.
  Cabozantinib: 60 mg QD orally in cycles of 28 days
- Metastatic or Unresectable Carcinoid: Patients were stratified by primary tumor site but received the same treatment. This cohort had advanced or metastatic carcinoid tumor.
  Cabozantinib: 60 mg QD orally in cycles of 28 days
Arm/Group | Metastatic or Unresectable PNET | Metastatic or Unresectable Carcinoid
All-Cause Mortality (participants affected / at risk) | 1/20 | 3/41
Serious Adverse Events (participants affected / at risk) | 15/20 | 24/41
Other Adverse Events (participants affected / at risk) | 20/20 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic or Unresectable PNET (N=20) | Metastatic or Unresectable Carcinoid (N=41)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Autoimmune disorder (Immune system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 3
Hypertension (Vascular disorders) | 1 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 5
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Lipase increased (Investigations) | 1 | 4
Lymphocyte count decreased (Investigations) | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pain (General disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Serum amylase increased (Investigations) | 0 | 2
Skin infection (Infections and infestations) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic or Unresectable PNET (N=20) | Metastatic or Unresectable Carcinoid (N=41)
Abdominal distension (Gastrointestinal disorders) | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 10 | 20
Activated partial thromboplastin time prolonged (Investigations) | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Akathisia (Nervous system disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 14 | 18
Alkaline phosphatase increased (Investigations) | 10 | 20
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 6
Anal hemorrhage (Gastrointestinal disorders) | 1 | 1
Anal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 11 | 23
Anorexia (Metabolism and nutrition disorders) | 10 | 12
Anxiety (Psychiatric disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 15 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 | 1
Blood antidiuretic hormone abnormal (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 4 | 2
Blurred vision (Eye disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chills (General disorders) | 2 | 0
Cholesterol high (Investigations) | 0 | 2
Cognitive disturbance (Nervous system disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 3
Conjunctivitis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Creatinine increased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Depression (Psychiatric disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 12 | 32
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 6
Dry eye (Eye disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 4 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 5
Dysgeusia (Nervous system disorders) | 2 | 15
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Dysphasia (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 6 | 10
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 1
Fatigue (General disorders) | 16 | 32
Fever (General disorders) | 5 | 2
Fibrinogen decreased (Investigations) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 5
Flushing (Vascular disorders) | 1 | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 6
Gum infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 5 | 6
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 0
Hot flashes (Vascular disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 29
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 8 | 20
Hyperthyroidism (Endocrine disorders) | 0 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 12
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 6
Hypokalemia (Metabolism and nutrition disorders) | 6 | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 8 | 16
Hyponatremia (Metabolism and nutrition disorders) | 6 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 14
Hypotension (Vascular disorders) | 1 | 2
Hypothyroidism (Endocrine disorders) | 4 | 9
INR increased (Investigations) | 1 | 5
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 | 0
Investigations - Other, specify (Investigations) | 3 | 10
Lip pain (Gastrointestinal disorders) | 1 | 0
Lipase increased (Investigations) | 3 | 10
Localized edema (General disorders) | 2 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 6
Memory impairment (Nervous system disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 7 | 12
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 12 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 2
Neutrophil count decreased (Investigations) | 4 | 10
Non-cardiac chest pain (General disorders) | 2 | 2
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 3 | 4
Pain (General disorders) | 8 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 8
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 9
Palpitations (Cardiac disorders) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Platelet count decreased (Investigations) | 9 | 17
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Prostate infection (Infections and infestations) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Serum amylase increased (Investigations) | 4 | 13
Sinus tachycardia (Cardiac disorders) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Stomach pain (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Tremor (Nervous system disorders) | 0 | 1
Urine discoloration (Renal and urinary disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 7
Weight loss (Investigations) | 4 | 9
White blood cell decreased (Investigations) | 7 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT01466036/Prot_SAP_000.pdf